CLINICAL TRIAL: NCT06686329
Title: Physical Activity to Prevent and Treat Hyperglycemia from a Mistimed Bolus Insulin Dose: the MISSED DOSE Study
Brief Title: Physical Activity to Prevent and Treat Hyperglycemia from a Mistimed Bolus Insulin Dose
Acronym: Missed Dose
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jane Yardley (Other)
Collaborators: Diabetes Québec (Other)
Responsible Party: Sponsor-Investigator, Jane Yardley, Research unit director, PhD, Institut de Recherches Cliniques de Montreal
Organization: Institut de Recherches Cliniques de Montreal (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-1288
Record Dates: First submitted 2024-11-06; First posted 2024-11-13 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2024-10

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1 diabetes; Exercise; Hyperglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity; Hyperglycemia | interventions — Walking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- All participants (Experimental): All participants will be in a single arm that undergoes three separate interventions. These interventions will include three different mealtime insulin administration: i) 15 minutes prior to eating, ii) post-prandially when alerted to rapidly rising glucose (increase of 0.2 mmol/L/min) or hyperglycemia (> 10.0 mmol/L) by CGM, and iii) the same conditions as ii) but with a 15-minute walk performed immediately after insulin administration.
  Interventions: Behavioral: Control (CON); Behavioral: Missed Dose (MISS); Behavioral: Missed Dose + 15min walk (MISS+EX)

INTERVENTIONS:
Behavioral: Control (CON) — Standardized meal with insulin administered 15 minutes before eating
Behavioral: Missed Dose (MISS) — Standardized meal with insulin administered post-prandially when alerted to rapidly rising glucose (increase of 0.2 mmol/L/min) or hyperglycemia (> 10.0 mmol/L) by CGM
Behavioral: Missed Dose + 15min walk (MISS+EX) — Standardized meal with insulin administered post-prandially when alerted to rapidly rising glucose (increase of 0.2 mmol/L/min) or hyperglycemia (> 10.0 mmol/L) by CGM with a 15-minute walk performed immediately after insulin administration

SUMMARY:
People living with type 1 diabetes (PwT1D) are recommended to administer insulin 10-15 minutes before meal consumption (pre-bolus), to account for the delay in the glucose lowering action associated with subcutaneously administered insulin. Due to the demands of day-to-day life, pre-bolusing is not always possible or may be forgotten. With continuous glucose monitors (CGMs), PwT1D may be alerted to this missed insulin dose by a CGM alert, including rapidly rising glucose (change >2.5mmol/L/15min) or hyperglycemia (>10.0 mmol/L), and deliver a mistimed (post-prandial) dose in response to CGM alert.

This study was designed to determine the effect of combining a post-prandial/mistimed insulin dose with 15 minutes of brisk walking. It is expected that walking will help to minimize or prevent hyperglycemia after a mistimed bolus insulin dose, as well as blunt the rise in glucose following a mistimed insulin dose.

DETAILED DESCRIPTION:
While important for managing glucose concentration, achieving consistent pre-prandial dosing is difficult. A recent study of 3,945 adults living with T1D found an average of six missed bolus doses during a 14-day period, with each missed dose being associated with -1.7% (-1.8, -1.6) less time in target range. An increase of 5% in time in range is a clinically significant improvement. The frequency of missed boluses reported by adolescents and young adults is especially high with 33% of those aged 13 - 18 years (n=1513), and 43% of those aged 18 - 26 years (n=1160) reporting more than one mistimed insulin delivery per week in a USA clinic registry cohort. Missing or mistiming two bolus doses weekly can raise HbA1c, a 3-month proxy of average glucose, by 0.5%. A 1% increase in HbA1c is associated with a 2.2- and 1.8-fold increase in the risk of developing nephropathy and retinopathy, respectively.

This large increase in HbA1c from just two missed or mistimed doses weekly is likely due to the subsequent duration and severity of hyperglycemia. Upon recognition of a mistimed insulin dose, blood glucose (BG) levels may already be rising rapidly or in a hyperglycemic range (>10.0 mmol/L) causing the duration of the resulting glucose excursion to be prolonged. Common explanations for missed doses include forgetting, disruption to usual routine (ex. travelling), dosing interfered with performing activities, hypoglycemia avoidance, injection pain, and embarrassment.

To meet the increased energy demands of PA, glucose uptake in contracting skeletal muscle increases through mechanisms which are dependent and independent of insulin. In the context of T1D this increased uptake can be problematic for maintaining normoglycemia because insulin-mediated glucose uptake does not decrease, as it does in people without diabetes. Additionally, PA decreases blood flow to the gut and slows gastric emptying which delays the entry of glucose into circulation following the consumption of food, and blunts the rise in blood glucose following food consumption in people without diabetes. While the glucose lowering effects of PA are generally problematic for people living with T1D due to an increased risk of hypoglycemia, PA could be useful to reduce glucose concentration when it is increasing rapidly, such as after a mistimed insulin dose. In the context of a mistimed insulin dose, PA may be beneficial as it: 1) begins to lower blood glucose concentration immediately independently of insulin, 2) increases sensitivity to insulin, and 3) delays glucose entry into circulation. Therefore, PA may be a useful strategy to lower blood glucose more quickly when combined with an insulin dose following recognition of a mistimed dose.

One study has investigated the effect of postprandial walking on the glucose concentration of people living with T1D and found that, compared to remaining sedentary after a meal, 15 minutes of brisk walking lead to a 36.2% and 47.2% reduction in peak glucose and incremental area under the curve (iAUC) of capillary glucose during the 2 hours after a meal, respectively. The exact timing of insulin dosage in the aforementioned study is unclear but occurred sometime within 10 minutes of the onset of meal consumption.

Pretest measures: Interested participants will be invited to the IRCM. Participants will be asked questions related to diabetes management, PA levels, and medication. Resting blood pressure and heart rate will also be measured. Where participants are eligible, anthropometric characteristics will be measured using standard protocols. Estimated A1c will be obtained with the last 30-days of CGM data. Participants will be asked to answer to some questionnaires about their barriers to physical activity, diabetes distress and socio-demographic characteristics. Those who meet all eligibility criteria and complete informed consent forms will be asked to test the standardized meal in order to determine the insulin bolus that will then be used during the three intervention visits. Participants will also perform an estimated maximal aerobic capacity test on a treadmill.

Testing sessions: Participants will be asked to arrive at the lab between 11am and 2pm on three occasions. This study will consist of three separate testing sessions where participants consume a standardized meal. Participants will administer their mealtime insulin bolus under three conditions: i) 15 minutes prior to eating (CON), ii) post-prandially when alerted to rapidly rising glucose (increase of 0.2 mmol/L/min) or hyperglycemia (> 10.0 mmol/L) by CGM (MISS), as well as iii) the same conditions as MISS but with a 15-minute walk performed immediately after insulin administration (MISS+EX).

Capillary blood glucose will be assessed every 30 minutes during the intervention visits. Participants will remain in the testing facility for 3 hours after the meal, provided that their CGM glucose has returned to target range (4.0-10.0 mmol/L). During the three hours after the meal, participants will not consume additional food (excluding hypoglycemia treatment), engage in physical activity, or administer additional correction insulin. Participants will be asked to match their daily food and insulin intake as closely as possible from one testing session to the next for the day before and during the morning before each intervention visit. Participants will be provided with log sheets to assist in this task and will also be asked to avoid strenuous exercise and alcohol intake the day before and the day of each intervention visit.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-24 years
* Type 1 diabetes diagnostic for at least two years
* Estimated glycated hemoglobin or glucose management indicator obtained from the past 30 days of CGM data of < 9.9%
* Use a Dexcom G7 CGM in routine care

Exclusion Criteria:

* Changes in insulin management strategy within the past 2 months
* Diagnosis of gastroparesis
* Having a condition that could render exercise harmful
* Intolerance to gluten and lactose
* Having significant renal disease (e.g., eGRF < 30 ml/min)
* Inability to provide informed consent due to cognitive deficit
* Currently taking other medications (other than insulin) that may alter glucose metabolism (e.g., non-insulin antihyperglycemic drugs such as sglt2-inhibitors, corticosteroids), unless dosages thereof have been stable for more than three months
* For women, being pregnant or breastfeeding

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Mean glucose | From 0 minute to 180 minutes
  Mean glucose, adjusted for baseline glucose, from the start of the meal until 3 hours after the meal

SECONDARY OUTCOMES:
Automated insulin | From 0 minute to 180 minutes
  Amount of insulin delivered by automated treatment systems during the three hours after the meal
Time in range | Up to 6 hours after the meal, up to 12 hours after the meal, overnight (midnight-6am) and up to 24 hours after the meal
  Time in range (4.0-10.0 mmol/L) over time periods of 6 hours, 12 hours, overnight (midnight-6am) and 24 hours after the meal to investigate any delayed or prolonged effects.
Time below range | Up to 6 hours after the meal, up to 12 hours after the meal, overnight (midnight-6am) and up to 24 hours after the meal
  Time below range (<4.0 mmol/L) over time periods of 6 hours, 12 hours, overnight (midnight-6am) and 24 hours after the meal to investigate any delayed or prolonged effects.
Time above range | Up to 6 hours after the meal, up to 12 hours after the meal, overnight (midnight-6am) and up to 24 hours after the meal
  Time above range (>10.0 mmol/L) over time periods of 6 hours, 12 hours, overnight (midnight-6am) and 24 hours after the meal to investigate any delayed or prolonged effects.
Area under the curve | Up to 6 hours after the meal, up to 12 hours after the meal, overnight (midnight-6am) and up to 24 hours after the meal
  Area under the curve (AUC) over time periods of 6 hours, 12 hours, overnight (midnight-6am) and 24 hours after the meal to investigate any delayed or prolonged effects.
Coefficient of variation | Up to 6 hours after the meal, up to 12 hours after the meal, overnight (midnight-6am) and up to 24 hours after the meal
  Coefficient of variation (CV%) over time periods of 6 hours, 12 hours, overnight (midnight-6am) and 24 hours after the meal to investigate any delayed or prolonged effects.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de recherches cliniques de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No